CLINICAL TRIAL: NCT01388257
Title: A National, Multicenter, Randomized Open-Label Study of Proctological Surgery Efficacy on Anoperineal Fistulas Healing in Crohn's Disease Patients Treated With Adalimumab. (Official French Title: "Étude Nationale, Multicentrique, randomisée et en Ouvert de l'efficacité de la Chirurgie Proctologique Sur la Cicatrisation Des Fistules anopérinéales de la Maladie de Crohn Chez Des Patients traités Par Adalimumab")
Brief Title: Anal Crohn Fistula Surgery
Acronym: FACC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: French Society of Coloproctology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNFCP-001
Record Dates: First submitted 2011-07-04; First posted 2011-07-06 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: Crohn Disease; Fistula; Anoperineal Fistula; Anal Fistula
Keywords: Crohn Disease; Anoperineal fistula; Anal fistula; Proctology; Drainage; Colorectal Surgery; Fistulotomy; Plug; Advancement flap; Glue; Anti Tumor Necrosis Factor-alpha; Adalimumab
MeSH Terms: conditions — Crohn Disease; Fistula; Rectal Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surgery (Experimental): Seton drain removal is associated with proctological surgery.
  Interventions: Procedure: All types of surgery procedures
- Simple seton drain removal (Other)
  Interventions: Procedure: Simple seton drain removal

INTERVENTIONS:
Procedure: All types of surgery procedures — All types of surgery procedures used for anoperineal fistula repair. Surgery procedures include fistulotomy, biological glue, rectal advancement flap and plug.
  Arms: Surgery
Procedure: Simple seton drain removal — Patients are simply followed after seton drain removal.
  Arms: Simple seton drain removal

SUMMARY:
The purpose of this study is to demonstrate, in patients treated with adalimumab, the efficacy of proctological surgery in anoperineal fistula healing after the removal of seton drain.

ELIGIBILITY:
Inclusion Criteria:

* male or female 18 years or older,
* women of childbearing age who use an effective contraception method or women incapable of becoming pregnant [(i.e. postmenopausal women for 1 year or surgically sterile (hysterectomy and/or bilateral oophorectomy)],
* Patient with fistulizing anoperineal Crohn's disease. Anoperineal fistulas can be associated with ileal, colic or rectal lesions,
* Patient with at least 1 anoperineal fistula drained with a seton for more than 1 month,
* Patient treated with adalimumab for more than 1 month,
* Patient who agrees to undergo surgery for its drained fistula(s),
* Patient with immunosuppressive therapy (azathioprine, 6-mercaptopurine ou methotrexate) stable for at least 3 months or patients without immunosuppressive therapy,
* Patient who gave signed written informed consent after having received verbal explanation and written information related to the trial.

Exclusion Criteria:

* Pregnant or breastfeeding women,
* Patient having a perineal abscess,
* Patient with a high anovaginal fistula that cannot be treated, according to the investigator ,with fistulotomy, gluing, biodegradable plug or advancement flap,
* Patient treated with a daily dose of corticosteroids of more than 20 mg (a dose of more than 20 mg daily will be authorized during the study),
* Contraindication to proctological surgery on the drained fistula(s),
* Patient presenting with somatic or psychic signs or symptoms that are not compatible with his/her participation in the trial according to the investigator,
* Patient who participate in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2011-10; Primary Completion 2016-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients having a clinical healing of their anoperineal fistulas in Crohn disease | 12 months after seton drain removal

SECONDARY OUTCOMES:
Proportion of patients having more than half of their fistulas healed | 3, 6, 12 and 24 months after seton drain removal
Change in Crohn disease activity assessed by Crohn's Disease Activity Index (CDAI) and Perianal Disease Activity Index (PDAI) | 3, 6, 12 and 24 months after seton drain removal
Change in anal continence assessed by Wexner and Vaizey scores | 12 and 24 months after seton drain removal
Crohn's Disease Endoscopic Index of Severity (CDEIS) | 12 months after seton drain removal
Change in patients' quality of life, assessed by the Inflammatory Bowel Disease Questionnaire (IBDQ) | 12 and 24 months after seton drain removal
Change in fistula activity assessed by magnetic resonance imaging (MRI) | 6, 12 and 24 months after seton drain removal
  Change in fistula activity assessed by MRI (Van Assche score and absence of contrast enhancement after injection of gadolinium with regards to fistulous tract
Change in discomfort and impact assessed by the patient using a visual analog scale (VAS) | 3, 6, 12 and 24 months after seton drain removal

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Abramowitz, MD, Principal Investigator — Hôpital Bichat-Claude Bernard
Locations (15):
- France (15):
  - CHU Bordeaux - Hôpital Saint André - Department of Hepato Gastroenterology, Bordeaux, Aquitaine
  - Maison de Santé Protestante de Bordeaux Bagatelle - Department of Proctology, Talence, Aquitaine
  - Clinique universitaire de chirurgie Digestive et de l'urgence, Hopital Universitaire Michallon - Colorectal Surgery Unit, Grenoble, Auvergne-Rhône-Alpes
  - CHU Pontchaillou - Department of Digestive Diseases, Rennes, Brittany Region
  - Polyclinique de Franche-Comté - Department of Proctological Surgery, Besançon, Franche-Comté
  - CHU de Rouen - Departement of Hepato Gastroenterologie and Nutrition, Rouen, Haute Normandie
  - Clinique des Cèdres - Hepato-Gastroenterology Department, Cornebarrieu, Midi-Pyrénées
  - Clinique Saint Jean Languedoc - Department of Gastroenterology, Toulouse, Midi-Pyrénées
  - Hôpital Nord de Marseille - Gastroenterology Department, Marseille
  - Hôpital de POISSY, Poissy
  - Polyclinique de l'Océan, Saint-Nazaire
  - Hôpital Louis Mourier - Department of Hepato-Gastroentérologie, Colombes, Île-de-France Region
  - Institut de Proctologie Léopold Bellan - Groupe Hospitalier Paris Saint Joseph - Department of Colo-Proctology, Paris, Île-de-France Region
  - Institut Mutualiste Montsouris - Proctology Unit, Paris, Île-de-France Region
  - Hôpital Bichat-Claude Bernard - Gastro-enterology Department, Paris, Île-de-France Region

REFERENCES:
- [Derived] Abramowitz L, Brochard C, Pigot F, Roumeguere P, Pillant H, Vinson Bonnet B, Faucheron JL, Senejoux A, Bonnaud G, Meurette G, Fayette JM, Train C, Staumont G, Siproudhis L, Bouchard D. Surgical closure, mainly with glue injection and anti-tumour necrosis factor alpha, in fistulizing perianal Crohn's disease: A multicentre randomized controlled trial. Colorectal Dis. 2022 Feb;24(2):210-219. doi: 10.1111/codi.15947. Epub 2021 Oct 23. PMID 34623746